CLINICAL TRIAL: NCT07367880
Title: The Monument Test : A New Tool for Assessing the Ability to Name and Identify Unique Entities. (TeDIMO)
Acronym: TeDIMO
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC25.0190_TeDIMO; 2025-A01292-47 (Other: ID RCB)
Record Dates: First submitted 2025-12-15; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer s Disease
Keywords: unique entities; denomination; identification; landmarks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People with Alzheimer Disease
  Interventions: Other: Identification and naming task
- Healthy elderly people
  Interventions: Other: Identification and naming task

INTERVENTIONS:
Other: Identification and naming task — Task of identification and naming of landmarks and celebrities

SUMMARY:
The goal of this study is to show a significant difference in performance between 2 groups of participants (healthy elderly people vs. people with Alzheimer Disease) in an identification and naming task involving famous monuments.

ELIGIBILITY:
Inclusion criteria :

* Alzheimer's disease:

  * Age ≥ 50 years and older
  * Possible or probable diagnosis of Alzheimer's disease according to the revised criteria of Mac Khann et al., 2011.
  * Score 18≤ MMSE ≤26
* Controls:

  * Age ≥ 50 years and older
  * MMSE score ≥ 26 For all subjects
  * No objection from the participant

Exclusion criteria

* Alzheimer's disease:

  * Persons referred to in Articles L1121-5 to L1121-8 of the CSP
* Controls:

  * Memory complaints
  * Persons referred to in Articles L1121-5 to L1121-8 of the CSP For all subjects
  * Significant neurological or psychiatric history
  * Taking psychotropic medication (neuroleptics)
  * Poor command of the French language, comprehension difficulties
  * Significant hearing or visual impairments (diplopia, nystagmus, scotoma, etc.)
  * Insufficient exposure to the media and/or socio-cultural knowledge (questionnaire) ; Deficit in face recognition (Benton Face Recognition Test)

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in the MA group will be selected from among patients attending memory consultations at the CMRR at the CHU Grenoble-Alpes (active file within the department) or from among patients referred to the CMRR by a doctor not practicing at the CMRR (general practitioners or specialists such as neurologists). Healthy elderly participants will be recruited from among those accompanying patients being monitored at the CMRR.
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2031-02-01 (Estimated); Study Completion 2032-02-01 (Estimated)

PRIMARY OUTCOMES:
Difference between the two groups in the identification and naming task involving famous landmarks | 1 month
  show a significant difference in performance between the two groups in the identification and naming task involving famous landmarks

SECONDARY OUTCOMES:
Development and standardization of a new tool for screening for naming disorders and visual identification of unique entities. | 5 years